CLINICAL TRIAL: NCT03897465
Title: Comparative Evaluation of the propertieS of the Contact LAyer Dressing LOMatuell Pro® Versus UrgoTul® in the Management of Acute Wounds
Brief Title: Lomatuell Pro® Versus UrgoTul® in the Management of Acute Wounds
Acronym: SLALOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lohmann & Rauscher (Industry)
Collaborators: RCTs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A02288-47
Record Dates: First submitted 2019-03-21; First posted 2019-04-01 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Acute Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lomatuell Pro (Experimental): Lomatuell Pro® is a wound contact layer consisting of wide-meshed tulle, impregnated with a polymer matrix, which form a gel on contact with wound exudate to facilitate moist wound healing.
  Interventions: Device: Lomatuell Pro
- UrgoTul (Active Comparator): UrgoTul® is a flexible contact layer with TLC (Technology Lipido-Colloid) healing matrix comprised of a conformable polyester mesh impregnated with hydrocolloid and petroleum jelly particles.
  Interventions: Device: UrgoTul

INTERVENTIONS:
Device: Lomatuell Pro — Patients will receive Lomatuell Pro dressings during 3 weeks. Lomatuell Pro® may be left in place up to 7 days; additional dressing changes can be performed as often as necessary according to the instruction for use.
  Arms: Lomatuell Pro
Device: UrgoTul — Patients will receive UrgoTul dressings during 3 weeks. UrgoTul® may be left in place up to 7 days; ; additional dressing changes can be performed as often as necessary according to the instruction for use.
  Arms: UrgoTul

SUMMARY:
Comparative evaluation of the propertieS of the contact LAyer dressing LOMatuell Pro® versus UrgoTul® in the management of acute wounds

DETAILED DESCRIPTION:
National, multicenter, prospective, randomized in parallel groups, non-inferiority, open-label investigation study.

ELIGIBILITY:
Inclusion Criteria:

* Acute wound: traumatic wound (dermabrasion, skin tears, other), small burns 1st and 2nd degree requiring the use of dressings
* Acute wound size between 3 cm² and 24 cm² (wound could be covered by 2 investigational products maximum)
* Wound whose duration is ≤ 3 days
* Both gender with an age ≥ 18 years
* Written confirmation from the study nurse that the patient was informed, orally agreed to participate and to comply with study treatment and planned visits
* Subject able to follow the protocol

Exclusion Criteria:

* Chronic and acute surgical wound
* Infected, moderately to strongly exudative and haemorrhagic wound
* Diagnosed underlying disease (e.g. diabetic neuropathy, stroke, etc.) which as judged by the investigator could interfere with the pain assessment
* Known allergy/hypersensitivity to any of the components of the investigational products
* Participation in other clinical investigation within one month prior to start of investigation
* Pregnant or breast-feeding women
* Person protected by a legal regime (tutorship or guardianship)
* Patients unable to manifest an oral consent to participate (e.g. dementia) or to understand the use of the VAS (visual analogue scale) tool
* Patient not covered by health insurance/social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2020-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daria TROFIMENKO, Study Director — Lohmann & Rauscher
Locations (1):
- CICA+, Limonest, France

REFERENCES:
- [Result] Meaume S, Kerihuel JC, Malatesta A, Roux F, Trofimenko D, Abel M. Non-inferiority randomised controlled trial of two contact layer dressings for the treatment of acute wounds (SLALOM). J Wound Care. 2025 Jul 2;34(7):496-505. doi: 10.12968/jowc.2024.0312. PMID 40632070

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on 11 February 2019. Last patient enrolled on 16 November 2020.
Period: Overall Study
Arm/Group | Lomatuell Pro | UrgoTul
Started | 78 | 81
Completed | 71 | 79
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — complete healing by V2 | 1 | 0
Not completed — occurence of exclusion criterion | 1 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- UrgoTul: UrgoTul® is a flexible contact layer with TLC healing matrix comprised of a conformable polyester mesh impregnated with hydrocolloid and petroleum jelly particles.
  UrgoTul: Patients will receive UrgoTul dressings during 3 weeks. UrgoTul® may be left in place up to 7 days; ; additional dressing changes can be performed as often as necessary according to the instruction for use.
- Total: Total of all reporting groups
Arm/Group | Lomatuell Pro | UrgoTul | Total
Number analyzed (Participants) | 78 | 81 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.83 (22.775) | 71.28 (22.364) | 72.53 (22.530)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 40 | 83
  Male | 35 | 41 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 78 | 81 | 159
Weight [Mean (Standard Deviation); unit: kg] — Population: Data missing for 2 patients
  kg
    number analyzed (Participants) | 78 | 79 | 157
    (all) | 67.85 (15.821) | 71.85 (14.362) | 69.86 (15.189)
Height [Mean (Standard Deviation); unit: cm] — Population: Data missing for 2 patients
  cm
    number analyzed (Participants) | 78 | 79 | 157
    (all) | 165.97 (10.198) | 167.82 (9.065) | 166.9 (9.658)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Data missing for 3 patients
  kg/m^2
    number analyzed (Participants) | 78 | 78 | 156
    (all) | 24.5 (5.07) | 25.5 (5.30) | 25.0 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Wound Dressing Changes Associated With a Pain <30 mm on Visual Analog Scale (VAS)
Description: To evaluate the main study objective, patients were asked to assess the pain they felt during the first dressing removal (D3±2 days) with a means of visual analog scale (VAS), a 100 mm straight line ranging from 0 to 100, where "0" refers to "no pain" and "100" to the "worst pain imaginable". The VAS score was directly measured by the investigator with a scale in millimetres and the number was entered in the patient's case report from (CRF).
Time Frame: At Visit 2 (Day 3 ± 2 days)
Measure: Number (95% Confidence Interval); unit: percentage of dressing changes
Arm/Group | Lomatuell Pro | UrgoTul
Number analyzed (Participants) | 77 | 81
percentage of dressing changes | 97.4 [97.01 to 98.06] | 97.5 [97.12 to 98.16]
Statistical Analysis 1: Comparison: Lomatuell Pro vs UrgoTul; Descriptive analysis of the primary endpoint was provided on per protocol population. The overall difference LomatuellPro (LP) - UrgoTul (UT) of the % of patients meeting main efficacy criterion was calculated with 95% bilateral confidence interval (CI). If lower limit of the 95% CI did not exceed the -10% value of pre-specified non-inferiority margin, non-inferiority had to be accepted. As a sensitivity analysis, the same analysis was performed on mITT (modified Intention-to-treat) population; Test type: Non-Inferiority — Pre-specified non-inferiority margin was 10%; Risk Difference (RD) = 1.4, 95% CI 2-sided [lower limit -10] (Upper Limit= +Infinity)

2. Secondary Outcome: Complete Healing
Description: Percentage of epithelialization of the wound at V3 calculated based on a blind assessment of wound photographs using W.H.A.T. assessment (W.H.A.T. = Wound Healing Analysing Tool is a program for assessment of the wound photos, which allows to obtain automatically-calculated results for wound area, wound dimensions, % of necrotic, granulation or epithelium tissues in the wound bed). "Complete healing" was defined as 100% of the wound area covered by the epithelium.
Time Frame: At Visit 3 (Day 21 or earlier, as soon as the wound is epithelialized)
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Lomatuell Pro | UrgoTul
Number analyzed (Participants) | 78 | 81
Participants | 48 | 55

ADVERSE EVENTS:
Time Frame: For each patient, adverse events were collected for maximum of 23 days from Baseline (D0) till the Final study visit (Day 21+2). There was no follow-up period in the study.
Description: Over the safety set (159 patients), 4 patients (2.5%) experienced an adverse event (AE) during the investigation: 3 patients from the LP group and 1 patient from the UT group. All the AEs were unexpected.
  All 3 AEs, registered in the LP group, were serious. The only AE, registered in the UT group, was non-serious.
  None of the registered (serious) adverse events were assessed as related to the study dressing or study procedure.
Arm/Group | Lomatuell Pro | UrgoTul
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/81
Serious Adverse Events (participants affected / at risk) | 3/78 | 0/81
Other Adverse Events (participants affected / at risk) | 0/78 | 1/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lomatuell Pro (N=78) | UrgoTul (N=81)
INFLAMED DIABETIC FOOT ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
NECROSIS DUE TO VASCULAR PROBLEM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
WORSENING OF THE WOUND (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lomatuell Pro (N=78) | UrgoTul (N=81)
Wound infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Open-label investigation design (nurses and patients knew which dressing was applied); Subjective pain scores assessment (by the patients).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT03897465/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT03897465/SAP_001.pdf